CLINICAL TRIAL: NCT01647685
Title: A Proof of Concept Study to Determine the Local Delivery and Efficacy of Intravenously Injected PEG-liposomal Prednisolone Sodium Phosphate (Nanocort) in Atherosclerotic Tissue in Subjects With Peripheral Artery Disease.
Brief Title: A Proof of Concept Study to Determine the Local Delivery and Efficacy of Nanocort
Acronym: DELIVER
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, E.S.stroes, Professor doctor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: NL39717.018.12
Record Dates: First submitted 2012-06-28; First posted 2012-07-23 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-05

CONDITIONS: Atherosclerosis
Keywords: Vesselwall inflammation; liposomal prednisolone
MeSH Terms: conditions — Atherosclerosis | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nanocort (Active Comparator): Two weekly IV infusions of 144 mg Nanocort (PEG-liposomal prednisolone sodium phosphate).
  Interventions: Drug: Nanocort
- Methylprednisolone (Active Comparator): Methylprednisolone sodium succinate 125 mg infusion.
  Interventions: Drug: Methylprednisolone
- Saline (Placebo Comparator): Saline solution (same solution brand as used to dilute/prepare Nanocort injection)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nanocort — Two weekly IV infusions of 150 mg Nanocort (PEG-liposomal prednisolone sodium phosphate).
  Other Names: Nanocort (PEG-liposomal prednisolone sodium phosphate).
  Arms: Nanocort
Drug: Methylprednisolone — Two weekly infusion iv methylprednisolone sodium succinate 125 mg infusion.
  Other Names: Methylprednisolone, Solu-medrol
  Arms: Methylprednisolone
Drug: Placebo — Saline solution (same solution brand as used to dilute/prepare Nanocort injection)
  Other Names: NaCl 0.9%
  Arms: Saline

SUMMARY:
A promising strategy to reduce CVD is to directly target inflammation at the level of the vessel wall. A potential drawback of anti-inflammatory strategies pertains to the thin line between inhibiting 'inappropriate' inflammation versus inducing immuno-suppression. One of the strategies to limit systemic immunosuppression is to strive for local delivery and prolonged efficacy and low systemic burden of the drug by encapsulating the compound in liposomes.

Liposome-encapsulated drugs efficiently target lesions and accumulate at a much higher extent at desired areas of interest. Thus, local delivery and prolonged efficacy can be very important tools to overcome the potential drawback anti-inflammatory drugs; namely an inappropriate immune suppression. In the present project, the investigators therefore aim to evaluate the delivery and superior efficacy of Nanocort above Prednison or placebo in patients with peripheral artery disease due to atherosclerosis. Because these patients will undergo an endarteriectomy the investigators will be able to collect atherosclerotic material after drug administration and thus evaluate the local delivery and compare the effects of Nanocort to Prednison or Placebo.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality in developed nations. CVD is primarily caused by atherosclerosis, a systemic disease characterized by lipid deposition in the subendothelial space with a concomitant, low-grade inflammatory reaction. Nowadays, most therapeutic interventions aimed at lowering CVD have thus far focused on modulating lipid levels, either lowering LDLc or increasing HDLc levels. Yet, since the introduction of statins 20 years ago, there have been few breakthroughs in the treatment of this disease. In fact, the recent failure of a potent HDL-increasing drug, i.e. torcetrapib, has emphasized the need to also consider non-lipid modulating targets.

A promising strategy to reduce CVD is to directly target inflammation at the level of the vessel wall. A potential drawback of anti-inflammatory strategies pertains to the thin line between inhibiting 'inappropriate' inflammation versus inducing immuno-suppression. One of the strategies to limit systemic immunosuppression is to strive for local delivery and prolonged efficacy and low systemic burden of the drug by encapsulating the compound in liposomes.

Liposome-encapsulated drugs efficiently target lesions and accumulate at a much higher extent at desired areas of interest. This approach is currently used for the clinical treatment of different types of cancer(liposomal doxorubicin) and fungal infections (liposomal amphotericine-B). Liposomes for other applications (rheumatoid arthritis, cystic fibrosis, multiple sclerosis and atherosclerosis) are being pre-clinically developed or investigated in clinical trials.

Recent pre-clinical studies in animal models corroborate that liposomal glucocorticoids effectively attenuate atherosclerotic plaque inflammation and exhibit improved pharmacokinetics and biodistribution. Also, local delivery through localization of liposomes at inflammatory sites and in local macrophages was demonstrated in animal models.

In humans, the potential of PEG-liposomes to target inflammatory sites has been showed by imaging of radioactive liposomes. However, the concept of local delivery and (prolonged) efficacy of liposomal corticosteroids at the inflammatory sites, such as atherosclerosis, and at local macrophages remains to be determined in humans.

Thus, local delivery and prolonged efficacy can be very important tools to overcome the potential drawback anti-inflammatory drugs; namely an inappropriate immune suppression. To proof this concept, the investigators need to evaluate the local delivery and efficacy at the site of inflammation (atherosclerosis) of intravenously administered liposomal glucocorticoids (Nanocort) compared to free glucocorticoids (Prednison). Only by comparing these two drugs, the investigators can prove the potential benefits of nanomedicine as a vehicle for local drug delivery. This can have major implications in future drug strategies for cardiovascular disease.

In the present project, the investigators therefore aim to evaluate the delivery and superior efficacy of Nanocort above Prednison or placebo in patients with peripheral artery disease due to atherosclerosis. Because these patients will undergo an endarteriectomy the investigators will be able to collect atherosclerotic material after drug administration and thus evaluate the local delivery and compare the effects of Nanocort to Prednison or Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria for study entry:

  1. Patients who are scheduled for endarterectomy due to peripheral artery disease.
  2. If using a statin, on stable therapy for at least 6 weeks prior to screening with no evidence of statin intolerance.
  3. For patients taking angiotensin-converting enzyme (ACE) inhibitors (ACE-I) or angiotensin-receptor blockers (ARBs), non-statin lipid-modifying therapy, thiazolidinediones, inhaled steroids, or leukotriene modifying agents, use of a stable dose for at least 6 weeks prior to baseline measurement.
  4. For patients taking Nonsteroidal anti-inflammatory drugs (NSAIDS), Cyclo-oxygenase-2 inhibitors (COXIBs), use of a stable dose for at least 6 weeks prior to baseline measurement.

Exclusion Criteria:

1. Current medical history of Auto-immune disease/vasculitis, active inflammatory diseases, proven or suspected bacterial infections. Recent (<1 month prior to screening) or ongoing serious infection requiring IV antibiotic therapy.
2. Recent or current treatment with medications that may have a significant effect on plaque inflammation, including but not limited to:

   * Steroids for at least 6 weeks prior to baseline measurement and during study (with the exception of inhaled steroids).
   * Biological based medicines (anti-TNF (ex. Infliximab), anti-IL-6 therapy (ex. Tocilizumab) or anti-IL-1 (ex. anakinra)) within 8 weeks before the baseline visit and during the study
   * No other Disease modifying antirheumatic drugs (DMRADS) within 6 weeks of baseline and during study (such as cyclosporine, azatioprine, etc.)
3. Known systemic disorder, such as hepatic, renal, hematologic or endocrine diseases, infections or malignancies, or any clinically significant medical condition that could interfere with the conduct of the study.
4. Subjects with a known ulcus ventriculi or duodeni.
5. Female subjects who are breastfeeding, pregnant or trying to get pregnant.
6. History of anaphylaxis, anaphylactoid (resembling anaphylaxis) reactions, or severe allergic responses.
7. History of hypersensitivity to methylprednisolone or any component of the formulation.
8. Any history of myopathy or a history of neuromuscular disorders (e.s, myasthenia gravis).
9. Any planned vaccinations.
10. Inability or unwillingness to comply with the protocol requirements, or deemed by investigator to be unfit for the study.
11. Subject has planned cardiac surgery, PCI or carotid stenting, or major non-cardiac surgery during the course of the study period or for 14 days after the last treatment.
12. Current medical history of drug or alcohol abuse within 12 months prior to screening.
13. Subjects are not permitted to enter the study if they have taken any investigational drug in the 3 months prior to study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Quantity of PEG liposomes in the atherosclerotic plaque and/ or in atherosclerotic macrophages as determined with a PEG antibody quantitative sandwich ELISA. | Participation of patient: maximally 12 days (infusion 1 on day-10 (+/-2days), infusion 2 on day-3, operation and sample collection on day 0) Data assessment: average 4 months.
  Quantity of PEG liposomes in the atherosclerotic plaque and/ or in atherosclerotic macrophages as determined with a PEG antibody quantitative sandwich ELISA.

SECONDARY OUTCOMES:
Differences between TNF-alpha levels in the supernatant of isolated macrophages from the atherosclerotic tissue as determined by quantitative sandwich ELISA | Participation of patient: maximally 12 days (infusion 1 on day-10 (+/-2days), infusion 2 on day-3, operation and sample collection on day 0) Data assessment: average 4 months.
  Differences between TNF-alpha levels in the supernatant of isolated macrophages from the atherosclerotic tissue as determined by quantitative sandwich ELISA
Concentration of corticosteroids in plaque. | Participation of patient: maximally 12 days (infusion 1 on day-10 (+/-2days), infusion 2 on day-3, operation and sample collection on day 0) Data assessment: average 4 months.
  Differences in concentration of corticosteroids in atherosclerotic plaque between 3 groups.

CONTACTS AND LOCATIONS:
Overall Officials: E S Stroes, MD PhD, Principal Investigator — AIDS Malignancy Consortium
Locations (1):
- AMC, Amsterdam, Amsterdam, Netherlands